CLINICAL TRIAL: NCT01659164
Title: Psychological Treatment for Attention-Deficit/Hyperactivity Disorder (ADHD) - Pilot Evaluation of a New Treatment Manual Based on CBT and DBT
Brief Title: Psychological Treatment for Adults With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Viktor Kaldo, Principal Investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012/333-31
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: ADHD
Keywords: Cognitive Behavioral Therapy; Dialectical Behavioral Therapy; Group Treatment; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group treatment (uncontrolled) (Experimental): Psychological treatment in group for adults with ADHD (pilot) during 14 weeks with focus on decreasing disabilities due to the condition.
  Interventions: Behavioral: Group treatment for adults with ADHD

INTERVENTIONS:
Behavioral: Group treatment for adults with ADHD — 14 weeks of group treatment for adults with ADHD

SUMMARY:
The purpose of this uncontrolled pilot study is to develop and make an initial evaluation of a new treatment manual for treatment of ADHD in adults. The objectives in the treatment is to build relational skills, skills in organizing and structuring everyday life, handle difficult emotions and impulses etc. The treatment will be in a group format and it is hypothesized that the psychological intervention will result in reduced ADHD symptoms and to decreased experience of stress and depressive symptoms. The uncontrolled design does not allow for any causal inferences from the results, this pilot study is primarily to be seen as a preparation before a subsequent RCT.

DETAILED DESCRIPTION:
Approximately one-third of children with ADHD continue to be fully symptomatic into adulthood and many of the remainders often retain some residual problems that require treatment. Thus ADHD is a prevalent and chronic disabling disorder. Drugs provide first line treatment for adults with ADHD but are not enough for everybody, while we still lack proper evidence for promising psychological treatment. In addition to core symptoms of ADHD including regulatory difficulties of attention, activity level and impulses, difficulties with emotional regulation are common.

Follow-up studies of adults with ADHD have shown that only a few patients were offered sufficient treatment and support after the neuropsychiatric assessment and testing. The majority of adults diagnosed with ADHD are offered pharmacological treatment (stimulant medication) as the sole treatment. However, stimulant medication is not effective for up to 20-50 percent of adults as they may not experience symptom reduction or they are unable to tolerate the medication.

Consequently, the possible benefits of identifying and treating individuals with ADHD are extensive. Treatment of ADHD is preferably multimodal, i.e. consisting of more than one intervention.

There has been limited research to date concerning psychosocial treatments for adult ADHD. Studies of cognitive behavioral therapy (CBT) and dialectical behavior therapy (DBT) show that structured short-term therapies are promising in reducing ADHD related symptoms and increasing life quality. Focus in the CBT treatment is to build skills, increasing and compensating for deficits in the executive functioning due to impairments of the frontal lobe. DBT combines change-oriented skills from CBT with acceptance-oriented skills and core mindfulness skills. DBT skills have been tried out and validated as a promising intervention package for adults with ADHD through the research of Steven Safren and Bernd Hesslinger.

The objective of the planned study is to evaluate a new manual for group treatment, with a combination of treatment methods from Safrens and Hesslingers evidence-based treatment manuals. The aim of the pilot project is to create a clinically effective combination of the different methods of treatment, with a high degree of understanding, acceptance, use and perceived usefulness of the patients undergoing treatment. Both qualitative and quantitative data about patients' perceptions and use of the different methods will be collected during and after treatment to increase knowledge of how treatments can be developed and combined in order to better match the needs of patients.

ELIGIBILITY:
Inclusion Criteria:

1. * Clinical diagnosis of AD/HD
2. * Age 18-65
3. 17 or more on the Adult ADHD Self Report Scale (ASRS v1.1)
4. Not medically treated for adhd symptoms, or medically treated with central stimulants or comparable substance since at least one month with no significant changes in dosage and where no change in medical treatment is anticipated during the study time frame for the participant.
5. No change in any other medical treatment is anticipated during the study time frame for the participant.
6. Participant are by investigators considered able to follow through the training protocol and take part in measures taken during the study time frame
7. The participant hasn´t used drugs the last 3 months.

   Exclusion Criteria:
8. Diagnosed substance abuse according to DSM-IV criteria within 3 months prior to screening. Earlier episodic substance abuse is not excluding
9. Co-existing psychiatric condition that investigators believe will unable the participant to follow through the training protocol and take part in measures taken during the study time frame.
10. IQ ≤70 according to a neuropsychological assessment
11. * Suicidality risk which is assessed during the first assessment interview.
12. Organic brain syndrome
13. Serious somatic condition which will unable the participant to participate (through the training protocol)or, is anticipated to have a negative impact on the treatment results
14. Autism spectrum disorder (severe)
15. Severe depression
16. Other current psychological treatment for AD/HD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change (from baseline) in ASRS- v 1.1 | 14 weeks (post)
  ADHD Self Report Scale (self rating)

SECONDARY OUTCOMES:
Change (from baseline) in ADHD Rating Scale | 14 weeks (post)
  ADHD Rating Scale - assessed by a clinician
Change (from baseline) in EQ-5D | 14 weeks (post)
  Euroqol - (self report) to measure general health and quality of life
Change (from baseline) in ISI | 14 weeks (post)
  Insomnia Severity Index - (self report) to measure insomnia symptoms
Change (from baseline) in PSS-4 | 14 weeks (post)
  Perceived Stress Scale - (self report) to measure level of stress in everyday life
Change (from baseline) in Sheehan Disability Scale | 14 weeks (post)
  Sheehan Disability Scale - (self report) to measure level of disability in everyday life
Change (from baseline) in MADRS-S | 14 weeks (post)
  Montgomery-Åsberg Depression Rating Scale - (self report) to measure level of depression
Change (from baseline) in DERS | 14 weeks (post)
  Difficulties of Emotion Regulation Scale - (self report)

OTHER OUTCOMES:
Treatment evaluation | 14 weeks (post)
  The investigators design own questions in order to evaluate how the participants have experienced the intervention regarding to knowledge, usage of the treatment methods and possible difficulties that they have experienced during treatment. Our aim is to use these evaluations to evolve and improve the quality of the treatment manual.

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Kaldo, Ph.D., Principal Investigator — Karolinska Institutet
Locations (1):
- Internetpsykiatrienheten, Psykiatri Sydväst, SLSO, Stockholm, Sweden